CLINICAL TRIAL: NCT01340261
Title: Registry: Pediatric Pain Rehabilitation Program
Brief Title: Pediatric Pain Rehabilitation Program
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Gerard A. Banez, Pediatric Psychologist, Director of Pediatric Pain Rehabilitation Program, The Cleveland Clinic
Other Study IDs: 07-099
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Pediatric Chronic Pain
Keywords: Pediatric; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Pain Rehab Patients
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires are completed at admission, discharge, 1-month, 6 month, and yearly follow-up.

SUMMARY:
The purpose of this study is to describe the demographic, medical, and psychological/behavioral characteristics of children and adolescent patients admitted to the Cleveland Clinic Children's Hospital's Pain Rehabilitation Program. The data will also be used to evaluate the clinical outcomes of patients admitted to the program as well as to examine the impact of various background factors on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted into the Cleveland Clinic Children's Hospital's Pain Rehabilitation Program

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants admitted to the Cleveland Clinic Children's Hospital's Pain Rehabilitation Program are eligible for enrollment in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2007-03; Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard A Banez, PhD, Principal Investigator — Cleveland Clinic Children's Hospital
Locations (1):
- Cleveland Clinic Children's Hospital for Rehabilitation, Cleveland, Ohio, United States

REFERENCES:
- See also: Related Info — http://my.clevelandclinic.org/childrens-hospital/specialties-services/therapy-rehab/pain-rehab.aspx